CLINICAL TRIAL: NCT05671952
Title: Multi-center Study on Reducing Postoperative Pulmonary Complications in Elderly Patients Based on Comprehensive Intervention System
Brief Title: Multi-center Study on Reducing Postoperative Pulmonary Complications in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Taihe Hospital (Other); Wuhan Central Hospital (Other); Shanxi Cardiovascular Hospital (Other); Qinghai People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPC20221203
Record Dates: First submitted 2023-01-02; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pulmonary Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Application of integrated intervention system programs
  Interventions: Other: Application of integrated intervention system programs
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Application of integrated intervention system programs — Application of integrated intervention system programs
  Arms: intervention group

SUMMARY:
The purpose of this study is to carry out demonstrative comprehensive intervention for elderly patients in several hospitals to observe whether it can reduce the incidence and mortality of perioperative pulmonary complications in elderly patients and improve their perioperative prognosis.

DETAILED DESCRIPTION:
This study investigated the incidence of postoperative pulmonary complications in various hospitals, and carried out demonstrative comprehensive intervention for elderly patients in several hospitals according to the comprehensive intervention system program of perioperative pulmonary complications, to observe whether the perioperative prognosis can be improved and the quality of life can be improved, thus verifying and optimizing the current evaluation system and intervention system, and providing evidence support for further extensive application.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 years or older
2. receiving invasive ventilation during general anesthesia for surgery

Exclusion Criteria:

1. preoperative mechanical ventilation
2. procedures related to a previous surgical complication
3. a second operation after surgery
4. organ transplantation
5. discharged within 24 hours after surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | within one week after surgery

SECONDARY OUTCOMES:
Postoperative pulmonary complications | 30 days after surgery